CLINICAL TRIAL: NCT05610488
Title: Intravitreal Faricimab in Diabetic Macular Edema With Limited Response to Aflibercept
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vista Klinik (Other)
Responsible Party: Principal Investigator, PD Dr. med. Katja Hatz, Head of clinical research and medical retina, Vista Klinik
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FarDME
Record Dates: First submitted 2022-10-27; First posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Diabetic Macular Edema
Keywords: DME; poor responder; aflibercept; faricimab
MeSH Terms: interventions — faricimab; Intravitreal Injections; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vabysmo (Faricimab) 6 mg (Experimental): Vabysmo (Faricimab) 6 mg solution for intravitreal injection All consenting, enrolled patients will receive an intravitreal injection of faricimab 6 mg at baseline (week 0), at week 4, 8, 12 (=4x loading) and each of the following treat and extend visits up to month 12.
  Interventions: Drug: FARICIMAB 6 Mg in 0.05 mL INTRAVITREAL INJECTION, SOLUTION [VABYSMO]

INTERVENTIONS:
Drug: FARICIMAB 6 Mg in 0.05 mL INTRAVITREAL INJECTION, SOLUTION [VABYSMO] — Intravitreal injection of faricimab 6 mg at baseline (week 0), at week 4, 8, 12 (=4x loading) and each of the following treat and extend visits
  Other Names: Vabysmo

SUMMARY:
Title: Intravitreal faricimab in diabetic macular edema with limited response to aflibercept

Purpose: The purpose of this investigator initiated study is to identify the effects of intravitreal faricimab on recurrence-free treatment intervals and morphological features in diabetic macular edema (DME) in which the Optical coherence tomography (OCT) guided treatment interval failed to be extended to 6 weeks intervals in a treat and extend regimen using aflibercept.

Objectives: The primary objective is to evaluate the proportion of patients with an increased maximum treatment interval with intravitreal faricimab (compared to previous 4-week interval under aflibercept) in an OCT guided treat and extend regimen at month 6 and 12. (for further outcome measures see section Objectives)

DETAILED DESCRIPTION:
Title: Intravitreal faricimab in diabetic macular edema with limited response to aflibercept

Study purpose: The purpose of this investigator initiated study is to identify the effects of intravitreal faricimab on recurrence-free treatment intervals and morphological features in diabetic macular edema (DME) in which the Optical coherence tomography (OCT) guided treatment interval failed to be extended to 6 weeks intervals in a treat and extend regimen using aflibercept.

Objectives: The primary objective is to evaluate the proportion of patients with an increased maximum treatment interval with intravitreal faricimab (compared to previous 4-week interval under aflibercept) in an OCT guided treat and extend regimen at month 6 and 12.

The secondary objectives are:

* The mean maximum treatment interval with intravitreal faricimab at month 6 and 12.
* The number of treatments applied during the 12 months study period.
* The mean change in BCVA (Best Corrected Visual Acuity) from baseline (=switch to faricimab) to month 6 and 12.
* To compare the mean BCVA at baseline (=switch to faricimab) and month 6/12 in patients with extended treatment intervals under faricimab.
* The mean change in CS (Contrast Sensitivity) from baseline (=switch to faricimab) to month 6 and 12.
* The mean change in AllEye index (metamorphopsia index) from baseline (=switch to faricimab) to month 6 and 12.
* The mean change in central retinal thickness as measured in the central ETDRS ( Early Treatment Diabetic Retinopathy Study) subfield from baseline (=switch to faricimab) to month 6 and 12.
* To compare the incidence of qualitative OCT features like intraretinal fluid, subretinal fluid, and hyperreflective foci between baseline (=switch to faricimab) and month 6 and 12.
* Percentage of patients achieving a dry retina at month 6 and 12.
* The mean changes in FAZ (foveal avascular zone) area and vessel density as measured by OCT-Angiography (OCTA) from baseline (=switch to faricimab) to month 6 and 12.
* The change in quality of life (VFQ-25 scores) from baseline to 6 and 12 months.
* To evaluate the safety and tolerability of up to 4weekly dosing of faricimab in DME by determining the rates of adverse events and serious adverse events at 6 and 12 month

Population: This outpatient study population will consist of a representative group of male and female patients ≥ 18 years of age suffering from DME with a treatment interval of 4 weeks under aflibercept. All patients are pre-treated with intravitreal aflibercept for at least 6 months in a treat and extend regimen. For In-/Exclusion criteria see section Eligibility.

Sample size will be 30. This is a pilot study investigating faricimab in pretreated aflibercept high demanders with DME using a real-life like treat and extend schema. So far this population has not been investigated with faricimab. In the context of recent market approval in Switzerland a timely start of the study to generate prospective data in this population with the highest treatment burden is recommended.

Measurements and Procedures:

All consenting, enrolled patients will receive an intravitreal injection of faricimab 6 mg at baseline (week 0), at week 4, 8, 12 (=4x loading) and each of the following treat and extend visits. From visit 4 (week 12) onwards extension of treatment intervals is possible 2-week-stepwise, e.g. 4, 6, 8 weeks etc. Starting at week 12 at each visit the next treat and extend interval (and so the exact date of the next visit) will be defined depending on the following criteria:

1. Presence of any DME activity including:

   - sub- and/or intraretinal fluid within the central ETDRS (Early Treatment Diabetic Retinopathy Study) subfield and/or ETDRS inner ring

   → new treatment interval = last treatment interval reduced by 2 weeks but minimum interval is 4 weeks, which means 4 weeks interval stays at 4 weeks, 6 weeks interval is reduced to 4 weeks etc
2. No signs of DME activity:

   → new treatment interval = last treatment interval plus 2 weeks
3. If there was 2 times a recurrence at a certain interval, in this patient the treatment interval stays at the 2 weeks lower interval.

Efficacy assessment at 3 months is within loading phase; for efficacy assessments after 6, 9 and 12 months a treat and extend visit which takes place within 2 weeks before/after (meaning 24±2 weeks, 36±2 weeks and 48±2 weeks, respectively) can replace an extra assessment visit as far as the required examinations are performed.

Efficacy assessments:

* Spectral-domain Optical coherence tomography (SD-OCT) at each study visit from baseline through month 12.
* Best corrected visual acuity (BCVA) measurements using the ETDRS-testing charts at a testing distance of 4m following ETDRS (Early Treatment Diabetic Retinopathy Study) refraction protocol at baseline, week 4, month 3, 6, 9 and 12.
* Contrast sensitivity measurement at baseline, week 4, month 3, 6, 9, 12.
* AllEye metamorphopsia measurement (self-test) at baseline and at each study visit from baseline through month 12.
* Swept-source OCT-Angiography at baseline, month 3, 6, 9, 12.
* Fluorescein angiography (FA) at baseline and month 12.
* Quality of life questionnaires VFQ-25 at baseline and month 6 and 12.

Other assessments:

* Ophthalmic examinations (slit lamp exam, fundus ophthalmo-scopy, Intraocular pressure (IOP) by applanation tonometry)
* Color fundus photography at baseline and month 12.
* Vital signs: heart rate (HR), blood pressure (BP)
* Adverse events (ocular and non-ocular)

Study Product / Intervention:

This study will include the following drug:

Investigational therapy

• Faricimab (Vabysmo®) 6 mg solution for intravitreal injection The drug is supplied as a sterile liquid for intravitreal injection in single-use glass vials (commercial product as approved in Switzerland).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age and documented diagnosis of diabetes mellitus (Type 1 or Type 2)
* Patients with diagnosis of diabetic macular edema (DME).
* Pre-treatment with intravitreal aflibercept in a treat and extend regimen and failing to be extended from the minimum interval of 4 weeks by two weeks to a 6-weeks interval without recurring DME activity or showing persisting DME activity in all visits under 4-weekly aflibercept treatment for at least 6 months.
* Patients who have a Best corrected Visual Acuity (BCVA) of at least 20/160 (letter score 40 letters) in the study eye using ETDRS (Early Treatment Diabetic Retinopathy Study) charts.
* Willing and able to give written informed consent according to legal requirements, and who have signed the consent form prior to initiation of any study procedure including withdrawal from exclusionary medications for the purpose of this study.
* Willing and able to comply with study procedures.
* For women of childbearing potential: agreement to remain abstinent or use acceptable contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 3 months after the final dose of study treatment

Exclusion Criteria:

* Treatment with panretinal photocoagulation or macular laser within 3 months prior to Day 1 to the study eye
* Any intraocular or periocular corticosteroid treatment within 6 months prior to Day 1 to the study eye
* Prior administration of intravitreal faricimab in either eye
* Active intraocular or periocular infection or active intraocular inflammation in the study eye
* Any history of ocular disease other than DME that may confound assessment of the macula/ affect central vision in the study eye
* History of uncontrolled glaucoma in the study eye (intraocular pressure ≥25 mmHg despite anti-glaucoma medication).
* Aphakia with absence of the posterior capsule in the study eye.
* Extracapsular extraction of cataract with phacoemulsification within three months preceding Baseline, or a history of post-operative complications within the last 12 months preceding Baseline in the study eye (uveitis, cyclitis, etc.).
* Use of other investigational drugs at the time of baseline, or within 30 days or 5 half- lives of baseline, whichever is longer (excluding vitamins and minerals).
* Previous violation of the posterior capsule in the study eye unless as a result of laser posterior capsulotomy in association with prior, posterior chamber intraocular lens implantation.
* Currently untreated diabetes mellitus or previously untreated patients who initiated oral or injectable anti-diabetic medication within 3 months prior to Day 1.
* Uncontrolled blood pressure (systolic value >180 mmHg and/or a diastolic value >100 mmHg while the patient is at rest)
* Currently pregnant or breastfeeding, or intend to become pregnant during the study.
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk for treatment complications.
* History of hypersensitivity or allergy to fluorescein.
* Inability to obtain Optical Coherence Tomography (OCT), Optical Coherence Tomography Angiography (OCTA), fundus photographs or fluorescein angiograms of sufficient quality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
maximum treatment interval with intravitreal faricimab at month 12. | 12 months
  maximum treatment interval with intravitreal faricimab at month 12.

SECONDARY OUTCOMES:
BCVA | 12 months
  Best corrected visual acuity (BCVA) in letters and BCVA change (letters) from baseline (=switch to faricimab) to month 12.
injection number | 12 months
  Number of faricimab intravitreal treatments applied during the 12 months study period.
metamorphopsia index | 12 months
  AllEye index (metamorphopsia index) and change of AllEye index from baseline to month 12. The AllEye index (between 0 and 100) is a measure for quantification of metamorphopsia; high values implicate less metamorphosia.
CRT (Central retinal thickness) | 12 months
  Central retinal thickness (CRT, in µm) as measured in the central ETDRS subfield Spectral-Domain Optical coherence tomography (SD-OCT) and change in CRT from baseline to month 12.
VFQ-25 Quality of Life Score | 12 months
  National Eye Institute Visual Function Questionnaire (VFQ-25) total and subscores (maximum 100 points) and their change from baseline to month 12. Higher scores implicate better quality of life.
Contrast acuity (CA) | 12 months
  Contrast acuity (CA) measured as the area under the log CS function (AULCSF) and its change from baseline (=switch to faricimab) to month 12.
Contrast Sensitivity (CS) threshold | 12 months
  Cutoff Spatial frequency (Cutoff SF) in cycles per degree (cpd) and its change from baseline (=switch to faricimab) to month 12.
Intraretinal fluid | 12 months
  Presence of intraretinal fluid (yes/no) as a qualitative SD-OCT feature within the central ETDRS subfield at month 12.
Subretinal fluid | 12 months
  Presence of subretinal fluid (yes/no) as a qualitative SD-OCT feature within the central ETDRS subfield at month 12.
Hyperreflective foci | 12 months
  Presence of hyperreflective foci (yes/no) as a qualitative SD-OCT feature within the central ETDRS subfield at month 12.
FAZ (foveal avascular zone) area | 12 months
  FAZ (foveal avascular zone) area (mm2) as measured by OCTangiography (OCTA) and its change from baseline to month 12.
Vessel density (VD) | 12 months
  Vessel density (VD) as measured by OCTangiography (OCTA) and its change from baseline to month 12. VD is expressed as the ratio (%) of the total vessel area to the total area of analyzed region.
Adverse events | 12 months
  Rates of adverse events and serious adverse events at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Katja Hatz, MD, Principal Investigator — Vista Augenklinik Binningen

IPD SHARING:
Plan to Share IPD: No
IPD share on special request